CLINICAL TRIAL: NCT01803009
Title: Patients' Opinions and Responses to the National Cancer Institute's Colorectal Cancer Risk Assessment Tool
Acronym: CRC-RAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Peter Schwartz, Associate Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1210009869
Record Dates: First submitted 2013-02-15; First posted 2013-03-04 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One arm (Experimental): View CRC RAT and view presentation regarding risk of advanced adenoma
  Interventions: Behavioral: Patient views NCI CRC RAT; Behavioral: View presentation regarding current chance of having an advanced adenoma

INTERVENTIONS:
Behavioral: Patient views NCI CRC RAT
Behavioral: View presentation regarding current chance of having an advanced adenoma

SUMMARY:
Little is known about the impact of risk assessment tools on decision-making by patients and clinicians. In particular, even though the NCI Colorectal Cancer Risk Assessment Tool is one of the most prominent risk assessment tools available, no study has quantified its usability or impact on decision-making or uptake of screening. In this study, we will measure patients' satisfaction with the NCI CRC RAT, their perception of its usability and helpfulness, and its impact on their decision-making and behavior. In addition, we will assess the impact of adding information about their chance of having an advanced adenoma.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years old
* No colonoscopy performed in last 10 years, sigmoidoscopy in last 5 years, or fecal occult blood testing (including FIT) in last 1 year.
* Appointment with healthcare practitioner in upcoming month or within the past six months at one of five Indiana University Health primary care sites.

Exclusion Criteria:

* Undergoing workup for signs or symptoms consistent with colon cancer, such as weight loss, iron-deficiency anemia, change in bowel habits, or rectal bleeding.
* Enrolled in "Trial of a Computer-Based Presentation of Quantitative Information about Colorectal Cancer Screening"; Dr. Schwartz's study that recently completed enrollment.
* Diagnosis with any of the following conditions: Ulcerative colitis, Crohn disease, Familial adenomatous polyposis (FAP), Hereditary Nonpolyposis Colorectal Cancer (HNPCC), Personal history of colorectal cancer or adenomatous polyp
* Inability to speak and read English

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Satisfaction with NCI CRC RAT | 1 day
  19 Likert-scale questions regarding usability of and satisfaction with the questions asked by the website to assess individual risk and the information provided
Perceived risk of developing CRC | 1 day
  Six Likert-scale questions regarding the subject's perceived risk of developing CRC in next 5 years, 10 years, and lifetime, and compared to others of same age and gender.
Intent to be screened within six months | 6 months
  Three multiple-choice questions regarding intent to be screened in next six months in general or with colonoscopy or stool testing. (Answer options: Definitely, Probably, Probably not, and Definitely not)
Stage of readiness to screen | 1 day
  Measure calculated from patient's answers on 5 multiple-choice or Likert-scale questions
Preferred CRC screening test | 1 day
  Answer on a single multiple choice question, offering options of colonoscopy, stool test, or other.

SECONDARY OUTCOMES:
Uptake of CRC screening | 6 months after intervention
  Phone call follow up and check of medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Peter H. Schwartz, MD, PhD, Principal Investigator — IU School of Medicine
Locations (1):
- Indiana University Health, Indianapolis, Indiana, United States